CLINICAL TRIAL: NCT04094155
Title: Retinal Vessel Analysis (rGA) at the Patient Bed in the Context of Non-traumatic Subarachnoid Haemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Gerrit Alexander Schubert, Head of Vascular Neurosurgery and Neurovascular Research, RWTH Aachen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-061
Record Dates: First submitted 2019-09-10; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Non-traumatic Subarachnoid Haemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retinal fundoscopy (Experimental): Retinal vascular analysis by retinal fundoscopy over a 3 week period in stationary patients after aneurysmatic subarachnoid hemorrhage
  Interventions: Diagnostic Test: retinal vascular analysis

INTERVENTIONS:
Diagnostic Test: retinal vascular analysis — Retinal fundoscopy over a 3 week period in stationary patients after aneurysmatic subarachnoid hemorrhage

SUMMARY:
A subarachnoid hemorrhage occurs in about 10 out of 100,000 people each year. This bleeding leads to irritation and constriction of blood vessels in the brain (vasospasm) in two out of three people affected within four to 21 days and thus to reduced blood flow. This can lead to a stroke and serious damage. In order to be able to diagnose and treat a constriction of the blood vessels at an early stage, there are various examination methods which, however, have various disadvantages such as radiation exposure of the patient, low sensitivity or high effort. Therefore, the prediction and timely therapy of vascular constrictions is currently only successful in a few cases before the reduced blood flow has already led to irreversible damage.

The aim of this study is to investigate whether the so-called retinal vascular analysis can be used in addition to previous standard examinations for the early detection of diseases of the cerebral blood circulation. This method has few side effects and has been successfully used for 50 years to examine the blood circulation in the eye.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient, age ≥ 18 years
* Inpatient stay in the clinic
* Written informed consent for participation in the study prior to beginning of treatment
* Written consent for further evaluation of the images and for the scientific publication of the study results
* Non-traumatic subarachnoid haemorrhage confirmed by computer tomography or magnetic resonance tomography or cerebrospinal fluid puncture (collection of nerve water from the lower part of the lumbar spine

Exclusion Criteria:

* Female or male patient < 18 years
* Pregnancy, Lactation
* Lack of written consent to participate in the study and to further evaluate the image material collected
* Known allergy to MS eye drops (active substance: phenylephrine/tropicamide
* Narrow chamber angle, narrow angle glaucoma, Terson syndrome (if it makes retinal vascular imaging impossible
* Persons in a dependency or employment relationship with the investigator
* Persons who are accommodated in a facility by judicial or administrative order
* Receipt and intake of a study drug within the last 30 days
* Supine position in bed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Progression of Delayed cortical ischemia | 21 days
  Delayed cortical ischemia as ischemia in cranial computer tomography or cranial magnetic resonance tomography that occurred later than 24 hours after admission to hospital

SECONDARY OUTCOMES:
Occurrence of delayed ischemic neurological deficit (DIND) | 21 days
Angiographic vasospasm | 7 days
  Occurence of an angiographic vasospasm measured by:
  * Digital subtraction angiography at day 7 +/- 2 days or
  * transcranial doppler sonography: flow increase >150 cm/s absolute or increase >50 cm/s within 24 h
Metabolic deficiency supply | 21 days
  Measured as change in lactate-pyruvate ratio in microdialysis
Metabolic deficiency supply | 21 days
  Measured as change in reduction in parenchymal oxygen partial pressure measurement
Relative underperfusion | 21 days
  Measured by Perfusion-Computer-Tomography
Objective degree of recovery | 3 Month
  Measured by Glasgow-Outcome-Scale; Scale by which patients who have experienced brain damage can be divided into 5 groups that allow to describe the degree of recovery in a standardized and objective manner (1: death; 2: vegetative condition, the patient is unresponsive. The higher cognitive functions are extinguished; 3: severe disability, the patient is conscious, but cannot cope with normal everyday activities without help; 4: moderate disability, the patient can live largely independently, but is not able to pursue a normal working life; 5: light to no handicap, the neurological, physical, and psychological deficits are so low that the patient can participate normally in social and economic activities)

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit A Schubert, Prof. Dr., Principal Investigator — Principal Investigator
Locations (1):
- Uniklinik RWTH Aachen, Klinik für Neurochirurgie, Aachen, Germany

REFERENCES:
- [Derived] Albanna W, Conzen C, Weiss M, Seyfried K, Kotliar K, Schmidt TP, Kuerten D, Hescheler J, Bruecken A, Schmidt-Trucksass A, Neumaier F, Wiesmann M, Clusmann H, Schubert GA. Non-invasive Assessment of Neurovascular Coupling After Aneurysmal Subarachnoid Hemorrhage: A Prospective Observational Trial Using Retinal Vessel Analysis. Front Neurol. 2021 Jun 14;12:690183. doi: 10.3389/fneur.2021.690183. eCollection 2021. PMID 34194387